CLINICAL TRIAL: NCT05748223
Title: The Effect of Mindfulness Meditation on Bispectral Index Monitoring, Physiological Findings and Cortisol Levels During Dental Implant Surgery: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Mindfulness Meditation During Dental Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cenk Haytac, Profesor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Cukurova U
Record Dates: First submitted 2023-02-03; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Mindfulness; Dental Implant
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Group (Experimental): The patients in this group received mindfulness meditation before dental implant surgery.
  Interventions: Other: Mindfulness Meditation
- Conventional Group (No Intervention): The patients in this group did not receive mindfulness meditation before dental implant surgery.

INTERVENTIONS:
Other: Mindfulness Meditation — Mindfulness meditation has been reported to produce beneficial effects on a number of psychiatric, functional somatic, and stress-related symptoms and has therefore increasingly been incorporated into psychotherapeutic programs
  Arms: Mindfulness Group

SUMMARY:
The aim of this pioneer study was to evaluate the efficacy (heart rate value, blood pressure, oxygen saturation, cortisol levels, BIS monitoring, patients' anxiety) of Mindfulness Meditation as a sedative technique during dental implant surgery.

DETAILED DESCRIPTION:
Since anxiety is a form of psychological stress, an increase in anxiety results in a surge in stress levels. The role of sedation in dental surgery cannot be overemphasised. The reduction in pain and anxiety eventually causes better cooperation and patients' satisfaction. Therefore, balancing anxiety and/or stress levels in patients would be useful to ensure patient safety during treatment.Therefore, the aim of this pioneer study was to evaluate the efficacy (heart rate value, blood pressure, oxygen saturation, cortisol levels, BIS monitoring, patients' anxiety) of Mindfulness Meditation as a sedative technique during dental implant surgery.

ELIGIBILITY:
. The inclusion criteria were:

* age between 25-65 years-old
* single tooth loss in the maxillary premolar-molar region with partial bone healing (type 3) or fully healed ridge type 4
* sufficient bony ridge for implant placement without the need for simultaneous bone grafting or sinus lift procedure
* no signs of acute oral infection,
* more than 2 mm of keratinized gingiva at the site of surgery
* periodontally healthy (or successfully treated) and otherwise healthy or had well-controlled systemic disease (ASA classification I, II).

Exclusion criteria were

* diabetes mellitus
* smoking
* pregnancy;
* diagnosis of anxiety disorders/psychiatric disorder/ depression and whether or not they were seeking any form of treatment for these conditions;
* poor oral hygiene (plaque control record > 30%);
* history of radiation therapy at head and neck area and chemotherapy; bony pathologies; history of soft tissue grafting at the prospective implant site

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Change of Bispectral Index (BIS) monitoring | Change from baseline to 5th, 10th, 15th, 20th, 25th and 30th minutes
  The level of sedation achieved by meditation was assessed with BIS device. BIS values range between 100 and 0 and give the clinicians objective information about the depth of sedation.

SECONDARY OUTCOMES:
Cortisol | At the baseline, immediately before and 5-minutes after surgery for both groups.
  The cortisol levels were biochemically evaluated
Blood pressure | Every 5-minutes starting from baseline until the end of surgery for both groups
  systolic and diastolic blood pressure (in mmHg) via vital signs monitor for both groups
arterial blood oxygen saturation | Every 5-minutes starting from baseline until the end of surgery for both groups
  in 'percentage %' via vital signs monitor for both groups
heart rate value | Every 5-minutes starting from baseline until the end of surgery for both groups
  in 'beats per minute' via vital signs monitor for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ucak Turer, Professor, Principal Investigator — Professor in Periodontology Department
Locations (1):
- Cukurova University Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No